CLINICAL TRIAL: NCT03119324
Title: Evaluation of the Efficacy of a New Low Level Laser Therapy (LLLT) Home Protocol in the Treatment of the Temporomandibular Joint Disorders Related Pain. A Randomized, Double Blind Placebo Controlled Clinical Trial
Brief Title: Low Level Laser Therapy in the Treatment of Temporomandibular Joint Disorders (TMJDs) Related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Umberto Romeo, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URomeo
Record Dates: First submitted 2017-03-03; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Biomodulation; LLLT; Temporomandibular Joint Disorders; Pain management
MeSH Terms: conditions — Temporomandibular Joint Disorders; Agnosia | interventions — Lasers, Semiconductor; Drug Therapy, Computer-Assisted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B-Cure® diode laser (Experimental): Thirty patients receiving LLLT by the B-Cure® diode laser (Good Energies, Haifa, Israel) 808nm low power device at 5 Joules/min, 250 milliWatts 15 KiloHertz for 8', (40 Joules each) in contact mode directly over the painful area, twice a day for 7 consecutive days.
  The laser must be placed directly over the painful area, after having cleaned it with a soft cotton socket to remove skin impurities that could interfere with therapeutic light absorption.
  The first application is performed at the Department of Oral Sciences of Sapienza University of Rome by a laser expert investigator and serves as instruction. The remnants must be performed by the patients themselves at home, once on the first day and twice a day in the following 6 days.
  Patients were instructed to perform the applications always at the same time.
  Interventions: Device: B-Cure® diode laser
- B-Cure® diode laser sham device (Placebo Comparator): Thirty patients that follows the same protocol of the SG but receive a B-Cure laser® sham device, seemingly identical to the effective one but devoid of main diode source.
  The laser must be placed directly over the painful area, after having cleaned it with a soft cotton socket to remove skin impurities that could interfere with therapeutic light absorption.
  The first application is performed at the Department of Oral Sciences of Sapienza University of Rome by a laser expert investigator and serves as instruction. The remnants must be performed by the patients themselves at home, once on the first day and twice a day in the following 6 days.
  Patients were instructed to perform the applications always at the same time.
  Interventions: Device: B-Cure® diode laser sham device
- Nimesulide Ratiopharm® and Flexiban® (Active Comparator): Thirty patients follows the conventional drug therapy protocol, of two non-consecutive cycles of 5 days of Non Steroidal Anti Inflammatory drug, Nimesulide Ratiopharm® (100 mg a day), interspersed with one 5 days cycle of Myorelaxant, Flexiban® (10 mg a day).
  From day 1 to 5, patients assumed 50mg of Nimesulide Ratiopharm®, twice a day; from 6th to 10th day they assumed 10mg of Flexiban® in single dose, from day 11 to 15 they assumed 50mg of Nimesulide Ratiopharm® twice a day.
  Patients were instructed to assume the therapy always at the same time
  Interventions: Drug: Nimesulide Ratiopharm® and Flexiban®

INTERVENTIONS:
Device: B-Cure® diode laser — B-Cure laser® (Good Energies, Haifa, Israel) 808nm diode laser application in contact mode over painful area twice a day for 7 consecutive days
  Other Names: Diode laser
  Arms: B-Cure® diode laser
Device: B-Cure® diode laser sham device — B-Cure laser® (Good Energies, Haifa, Israel) application by sham device twice a day for 7 consecutive days
  Other Names: Sham device
  Arms: B-Cure® diode laser sham device
Drug: Nimesulide Ratiopharm® and Flexiban® — Five consecutive days assumption of Non Steroidal Anti Inflammatory drug, Nimesulide Ratiopharm® 50mg twice a day, followed by five consecutive days assumption of Myorelaxant, Flexiban®, 10mg once a day, followed by five consecutive days assumption of 50mg of Non Steroidal Anti Inflammatory drug, Nimesulide Ratiopharm®, twice a day
  Other Names: Drug protocol
  Arms: Nimesulide Ratiopharm® and Flexiban®

SUMMARY:
The Low Level Laser Therapy (LLLT) has been recently introduced with success in the management of the pain associated to this condition. This double blind placebo controlled clinical trial analyzes a new home LLLT protocol to verify whether it was possible to avoid to the repeated presence at dental chair required by traditional LLLT protocols.

DETAILED DESCRIPTION:
90 patients with pain deriving from mono- or bi-lateral TMJDs were enrolled in the study. Randomly subdivided in 3 groups. The Study Group (SG n=30) receive a LLLT by the B-cure Dental Pro 808nm diode low level laser (Biocare Enterprise Ltd, Good Energies, Haifa, IL). The therapeutic protocol previews 2 applications a day for 7 consecutive days performed at 5 Joules/min, 250 milliWatts and 15 KiloHertz for 8', (40 Joules total each) in contact mode over the painful area.

The first application is performed at the Department of Oral Sciences of Sapienza University of Rome, by a laser expert blinded examiner and serves as instruction. The remnants applications must be performed at home by the patients themselves.

The Placebo Group (PG n=30) follows the same protocol by a sham device, seemingly identical to the effective ones, including the pointer light, but devoid of the main diode source.

The Drug Control Group (DG n=30) follows the conventional drug treatment for TMJDs related pain, 2 non-consecutive cycles of 5 days of nimesulide (100mg a day), interspersed with one 5 days cycle of cyclobenzaprine hydrochloride (10 mg a day) Two pain evaluation are registered, before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* TMJD diagnosed clinically and by CT and MRI; presence of pain in the TMJ area or radiating to the face, jaw, or neck; reduced mouth opening or jaw locks, painful clicking, popping or grating when opening or closing mouth, occlusal alterations

Exclusion Criteria:

* Muscle tenderness; NSAIDs assumption within 3 weeks before the treatment; pregnancy; neurocognitive diseases; autoimmune diseases; connective diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Pain reduction laser groups | 7 days
  Pain assessment by the visual analogue scale (VAS) from Baseline, at day 1 before the treatment, and at day 7, after one week of laser protocol
Pain reduction drug control | 15 days
  Pain assessment by the visual analogue scale (VAS) from Baseline, at day 1 before the treatment and at day 15, after two weeks of drug assumption

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Romeo, Professor, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No